CLINICAL TRIAL: NCT05347602
Title: A Clinical Study to Evaluate the Safety and Efficacy of Microscopic Doses Oral Administration of Gold Nanoparticles (AuNPs) on Knee Joint Health and Function
Brief Title: Gold Factor on Knee Joint Health and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 4Life Research, LLC (Industry)
Collaborators: Professional Athletic Orthopedics (Unknown); St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GF-AuKHC46
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Knee Arthritis; Knee Osteoarthritis; Knee Pain Chronic; Knee Discomfort; Rheumatoid Arthritis; Knee Pain Swelling
Keywords: Knee joint health; Arthritis; Gold nanoparticles (AuNPs); Knee joint function; Osteoarthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid; Arthritis; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Fifty-one (51) subjects were determined eligible for the study after the screenings and then were divided into two groups, AuNP Supplement (n=26) and Placebo (n=25). The study was partially double-blinded, and divided into three phases as follows:
  Phase 1: Supplement and Placebo groups ingested Supplement and Placebo as instructed. This phase was double-blinded.
  Phase 2: Both groups underwent a month-long "wash out" period, during which they did not ingest any of the Supplement or Placebo. This phase was not double-blinded as all participants and the researchers were aware of the wash-out procedure.
  Phase 3: Both groups took the Supplement as instructed. This phase was open labeled, as all participants and the researchers were aware that all participants were ingesting the Supplement.
Who Masked: Participant, Investigator
Masking Description: Phase 1 was double-blinded, neither investigator nor participants know what products each participant was taking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1: double-blinded placebo-controlled Supplement vs Placebo (Other): Phase 1 (8 weeks): Supplement and Placebo groups ingested 3 oz of Supplement and Placebo per day respectively for the first four weeks as a loading dose, and then switched to 2 oz per day for weeks 5 - 8. This phase was double-blinded.
  Interventions: Dietary Supplement: Gold Factor (Gold Nanoparticles, AuNPs); Dietary Supplement: Placebo
- Washout Phase (No Intervention): Phase 2 (4 weeks): Both groups underwent a month-long "wash out" period, during which they did not ingest any of the Supplement or Placebo. This lasted from weeks 9-12. This phase was not double-blinded as all participants and the researchers were aware of the wash-out procedure.
- Phase 3: Supplement (Active Comparator): Phase 3 (8 weeks): Both groups took the Supplement at 3 oz per day as a loading dose for four weeks (weeks 13 - 16), and then 2 oz per day for the final four weeks (weeks 17 - 20). This phase was open labeled, as all participants and the researchers were aware that all participants were ingesting the Supplement.
  Interventions: Dietary Supplement: Gold Factor (Gold Nanoparticles, AuNPs)

INTERVENTIONS:
Dietary Supplement: Gold Factor (Gold Nanoparticles, AuNPs) — AuNP used in the study is an aqueous suspension of clean-surfaced, faceted gold nanoparticles that have extraordinary catalytic capabilities. AuNP were 8 - 28 nm in diameter, with varying shapes from bipyramids to polyhedrons. To avoid contamination, AuNP was suspended in ultra-pure water, and were not coated with any proteins or molecules to avoid negative reactions within living tissues. This resulted in a rose-pink color due to the incident light inducing a specific resonance known as the localized surface plasmon resonance. The AuNP supplement used in this study contains elemental gold at 6 ppm. Study dosage is 1 oz per day, which is about 0.17 mg elemental gold per day.
  Other Names: AuNP Supplement
  Arms: Phase 1: double-blinded placebo-controlled Supplement vs Placebo; Phase 3: Supplement
Dietary Supplement: Placebo — For the Placebo, water and red dye were mixed to create a placebo liquid with the same rose-pink shade as the AuNP supplement, along with flavoring that matched the AuNP supplement.
  Arms: Phase 1: double-blinded placebo-controlled Supplement vs Placebo

SUMMARY:
The purpose of this clinical study was to determine whether gold nanoparticles (AuNP) supplement holds clinical value in improving joint health, function, and quality of life for arthritis patients.

DETAILED DESCRIPTION:
The purpose of this clinical study was to determine whether gold nanoparticles (AuNP) supplement holds clinical value in improving knee joint health, function, and quality of life for arthritis patients. A total of 51 participants were followed for 20 weeks through a three phase longitudinal study. Both subjective and objective parameters were used to measure and monitor changes in knee joint health and function, as well as quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and <87 years of age
* Having arthritis
* Suffering from chronic knee pain
* Failed treatments to date - including surgery, Physical Therapy, NSAIDs
* Must agree to maintain the same eating, exercise, and sleep arrangements for the whole duration of the study

Exclusion Criteria:

* Having bacterial, intra-articular, or knee infections
* Had any knee related partial or complete total knee replacement within 3 months prior to the start of the study
* Had recent (3 months prior to start of the study) knee injection
* Currently on NSAIDs
* currently pregnant or lactating

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS): Pain score | 20 weeks
  The KOOS survey was chosen due to its repeatability, and it gave scores of 0-100 for four separate categories: Symptoms, Pain, Function & Daily Living, Sports & Recreational Activities, and Quality of Life. Under KOOS scoring guidelines, a score of zero represents extreme knee problems, and 100 represents complete function of the knee with no pain, discomfort, or other joint related problems.
Knee injury and Osteoarthritis Outcome Score (KOOS): Symptoms score | 20 weeks
  The KOOS survey was chosen due to its repeatability, and it gave scores of 0-100 for four separate categories: Symptoms, Pain, Function & Daily Living, Sports & Recreational Activities, and Quality of Life. Under KOOS scoring guidelines, a score of zero represents extreme knee problems, and 100 represents complete function of the knee with no pain, discomfort, or other joint related problems.
Knee injury and Osteoarthritis Outcome Score (KOOS): Function in Activities of Daily Living (ADL) score | 20 weeks
  The KOOS survey was chosen due to its repeatability, and it gave scores of 0-100 for four separate categories: Symptoms, Pain, Function & Daily Living, Sports & Recreational Activities, and Quality of Life. Under KOOS scoring guidelines, a score of zero represents extreme knee problems, and 100 represents complete function of the knee with no pain, discomfort, or other joint related problems.
Knee injury and Osteoarthritis Outcome Score (KOOS): Function in Sports and Recreation score | 20 weeks
  The KOOS survey was chosen due to its repeatability, and it gave scores of 0-100 for four separate categories: Symptoms, Pain, Function & Daily Living, Sports & Recreational Activities, and Quality of Life. Under KOOS scoring guidelines, a score of zero represents extreme knee problems, and 100 represents complete function of the knee with no pain, discomfort, or other joint related problems.
Knee injury and Osteoarthritis Outcome Score (KOOS): Quality of Life score | 20 weeks
  The KOOS survey was chosen due to its repeatability, and it gave scores of 0-100 for four separate categories: Symptoms, Pain, Function & Daily Living, Sports & Recreational Activities, and Quality of Life. Under KOOS scoring guidelines, a score of zero represents extreme knee problems, and 100 represents complete function of the knee with no pain, discomfort, or other joint related problems.
C-Reactive Protein | 20 weeks
  C-Reactive Protein levels were measured at T0 for baseline scores, and then measured again at T1, T2, and T3. As CRP levels are biomarkers of systemic inflammation, it was expected to see a decrease in CRP levels when taking AuNP Supplement.
Range of Motion Bilateral Flexion score | 20 weeks
  All participants completed a physical assessment conducted by an assigned physical therapist: Range of Motion Bilateral Flexion, Leg Press, Walk Test, Sit-to Stand and Single Leg Squats.
Leg Press repetition number | 20 weeks
  All participants completed a physical assessment conducted by an assigned physical therapist: Range of Motion Bilateral Flexion, Leg Press, Walk Test, Sit-to Stand and Single Leg Squats.
6-minute Walk distance (meter) | 20 weeks
  All participants completed a physical assessment conducted by an assigned physical therapist: Range of Motion Bilateral Flexion, Leg Press, Walk Test, Sit-to Stand and Single Leg Squats.
Sit-to Stand repetition number | 20 weeks
  All participants completed a physical assessment conducted by an assigned physical therapist: Range of Motion Bilateral Flexion, Leg Press, Walk Test, Sit-to Stand and Single Leg Squats.
Single Leg Squats repetition number | 20 weeks
  All participants completed a physical assessment conducted by an assigned physical therapist: Range of Motion Bilateral Flexion, Leg Press, Walk Test, Sit-to Stand and Single Leg Squats.

SECONDARY OUTCOMES:
Number of Event for Loss of Balance (LOB) | 20 weeks
  DorsaVi Assessments: Loss of Balance (LOB), Movement efficiency index, Squat Lumbar Flexion Deviation, Squat Lateral Shift Deviations, single leg squat scores, speed, and tibial inclination
Movement efficiency index | 20 weeks
  DorsaVi Assessments: Loss of Balance (LOB), Movement efficiency index, Squat Lumbar Flexion Deviation, Squat Lateral Shift Deviations, single leg squat scores, speed, and tibial inclination
Squat Lumbar Flexion Deviation score | 20 weeks
  DorsaVi Assessments: Loss of Balance (LOB), Movement efficiency index, Squat Lumbar Flexion Deviation, Squat Lateral Shift Deviations, single leg squat scores, speed, and tibial inclination
Squat Lateral Shift Deviation score | 20 weeks
  DorsaVi Assessments: Loss of Balance (LOB), Movement efficiency index, Squat Lumbar Flexion Deviation, Squat Lateral Shift Deviations, single leg squat scores, speed, and tibial inclination
single leg squat speed | 20 weeks
  DorsaVi Assessments: Loss of Balance (LOB), Movement efficiency index, Squat Lumbar Flexion Deviation, Squat Lateral Shift Deviations, single leg squat scores, speed, and tibial inclination
single leg squat tibial inclination | 20 weeks
  DorsaVi Assessments: Loss of Balance (LOB), Movement efficiency index, Squat Lumbar Flexion Deviation, Squat Lateral Shift Deviations, single leg squat scores, speed, and tibial inclination
Percentage of participants that would continue taking the product after the study ended. | 20 weeks
  Acceptability of AuNP Supplement was analyzed at the end of the study. Participants were asked if they would continue taking the product after the study in their final exit survey.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Lehman, MD, Principal Investigator — Professional Athletic Orthopedics
Locations (1):
- Professional Athletic Orthopedics, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No